CLINICAL TRIAL: NCT02936076
Title: Exercise as a Buffer Against Stress-induced Overeating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 592916-14; K01DK100498 (NIH)
Record Dates: First submitted 2016-10-13; First posted 2016-10-18 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise condition (Active Comparator): Participants randomized to the exercise condition will participate in a 12-week exercise training program. The exercise intervention will consist of both supervised and unsupervised exercise sessions and progress to 200 minutes/week of moderate-intensity exercise. Exercise bouts will be spread across 4-6 days and be at least 20 minutes in duration. During supervised visits, heart rate will be monitored by a member of the research staff to ensure that exercise is within the prescribed intensity range and ratings of perceived exertion and feeling state will be assessed periodically. Unsupervised exercise will be verified using objective physical activity monitors.
  Interventions: Other: Exercise intervention
- Delayed exercise condition (Placebo Comparator): Participants randomized to the delayed exercise condition will be asked not to change their exercise or eating habits over the 12-week period and will complete the same assessment measures as the exercise condition. However, following the completion of the 12-week period, participants will be given two options: 1) receive a one-on-one session with an exercise physiologist at our center and receive a written exercise program, and at this time point all study obligations will be completed, or 2) complete the identical exercise protocol as the 'exercise' condition.
  Interventions: Other: Delayed exercise intervention

INTERVENTIONS:
Other: Exercise intervention
  Arms: Exercise condition
Other: Delayed exercise intervention
  Arms: Delayed exercise condition

SUMMARY:
The purpose of this study is to examine the psychological benefits of chronic exercise as well as the effects of exercise training on eating behaviors and stress-induced overeating in overweight and obese women. Participants will be randomized to an 12-week exercise condition or a delayed exercise condition. Assessments will occur at baseline, 6 weeks, and 12 weeks and will include answering surveys in real-time using smartphones, several assessments of eating behaviors and dietary intake, and questionnaire measures of factors which could mediate the relationship between exercise and eating. Participants will be compensated for completing assessments and for adherence to the exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-60 years of age
* BMI 25 to <40 kg/m2
* Physically inactive (<60 min/week of physical activity)
* Must own a smartphone
* Must be willing to receive and respond to text message prompts for 14 days at baseline, 6 and 12 weeks

Exclusion Criteria:

* Shift workers
* Individuals who do not endorse stress-eating
* Recent weight loss or current enrollment in a weight loss program
* Women who are pregnant or plan on becoming pregnant in the next 6 months
* Any medical condition that would limit participation in physical activity
* Diabetes
* Inability to walk without an assisted device
* Inability to meet exercise recommendations
* Failure to adequately complete all baseline assessment measures

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Unick JL, Dunsiger SI, Leblond T, Hahn K, Thomas JG, Abrantes AM, Stroud LR, Wing RR. Randomized Trial Examining the Effect of a 12-wk Exercise Program on Hedonic Eating. Med Sci Sports Exerc. 2021 Aug 1;53(8):1638-1647. doi: 10.1249/MSS.0000000000002619. PMID 34261994

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise Condition: Participants randomized to the exercise condition will participate in a 12-week exercise training program. The exercise intervention will consist of both supervised and unsupervised exercise sessions and progress to 200 minutes/week of moderate-intensity exercise. Exercise bouts will be spread across 4-6 days and be at least 20 minutes in duration. During supervised visits, heart rate will be monitored by a member of the research staff to ensure that exercise is within the prescribed intensity range and ratings of perceived exertion and feeling state will be assessed periodically. Unsupervised exercise will be verified using objective physical activity monitors.
  Exercise intervention
- Delayed Exercise Condition: Participants randomized to the delayed exercise condition will be asked not to change their exercise or eating habits over the 12-week period and will complete the same assessment measures as the exercise condition. However, following the completion of the 12-week period, participants will be given two options: 1) receive a one-on-one session with an exercise physiologist at our center and receive a written exercise program, and at this time point all study obligations will be completed, or 2) complete the identical exercise protocol as the 'exercise' condition.
  Delayed exercise intervention
Period: Overall Study
Arm/Group | Exercise Condition | Delayed Exercise Condition
Started | 25 | 24
Completed | 19 | 20
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Condition | Delayed Exercise Condition | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (11.7) | 41.0 (10.0) | 40.4 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 22 | 22 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 4 | 4
  White | 21 | 16 | 37
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Stress-induced Overeating Measured Via Smartphone Surveys
Description: Participants completed EMA surveys (5x/day for 14 days). At each prompt they were asked if an eating episode occurred. If they indicated 'yes', they were asked to check all that apply: a) I ate past the point of feeling full, b) I ate more than usual, c) I had unplanned eating (i.e., consumed food when I don't usually eat and was not making up for a missed meal, or d) None of the above. If the participant responded with a, b, or c, it was classified as an 'overeating episode'. Further, at each prompt, participants were asked to the respond to the following: 'Right now I feel stressed' (1=not at all, 7=very much so). If the stress score was >=5 at the prompt just prior to an overeating episode, then it was considered a 'stress-induced overeating episode'.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Exercise Condition | Delayed Exercise Condition
Number analyzed (Participants) | 19 | 20
episodes | 0.74 (1.56) | 0.55 (1.0)

2. Primary Outcome: Percentage of Overeating Episodes Characterized as 'Overeating'
Description: If an eating episode occurred, participants were asked to check all that apply: a) I ate past the point of feeling full, b) I ate more than usual, c) I had unplanned eating (i.e., consumed food when I don't usually eat and was not making up for a missed meal, or d) None of the above. If response was a, b, or c, it was classified as an 'overeating episode'.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: % of eating episodes
Arm/Group | Exercise Condition | Delayed Exercise Condition
Number analyzed (Participants) | 19 | 20
% of eating episodes | 21.98 (3.32) | 26.62 (3.58)

3. Secondary Outcome: Change in Body Weight (% Initial Weight)
Description: Percent weight change from baseline to 12 weeks
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Exercise Condition | Delayed Exercise Condition
Number analyzed (Participants) | 19 | 20
percent change | -1.1 (3.5) | 0.4 (2.0)

4. Secondary Outcome: Stress as Measured Via Questionnaire
Description: The 10-item Perceived Stress Scale (Cohen 1988) was used to assess changes in stress by treatment arm from baseline to 12 weeks. Scores on this measure range from 0-40 with a higher score indicating greater perceived stress. Presented values are 12 week scores adjusted for baseline values.
Time Frame: Baseline and 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Exercise Condition | Delayed Exercise Condition
Number analyzed (Participants) | 19 | 20
units on a scale | 22.7 (0.8) | 21.5 (0.8)

ADVERSE EVENTS:
Time Frame: 12 weeks post randomization
Arm/Group | Exercise Condition | Delayed Exercise Condition
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02936076/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-11): https://cdn.clinicaltrials.gov/large-docs/76/NCT02936076/SAP_001.pdf